CLINICAL TRIAL: NCT04051411
Title: The Effects of Degenerative Mitral Regurgitation on Cardiac Structure and Function, Symptoms, and Exercise Capacity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Seth Uretsky, Medical Director, Cardiovascular Imaging, Atlantic Health System
Other Study IDs: 1444724
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; echocardiography; MRI
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current American College of Cardiology/American Heart Association guidelines recommend that patients with severe degenerative mitral regurgitation be considered for mitral valve surgery. There remains a debate within the cardiology community regarding the appropriate management of patients who remain asymptomatic. In this study the investigators will perform longitudinal follow-up data with cardiac MRI to inform the prophylactic surgery vs. close follow-up debate and to better define the natural history of this condition. The investigators hypothesize, that in the majority of patients mitral regurgitation will not worsen overtime, left ventricular hemodynamics will remain stable, exercise capacity will not decline, and symptoms will not worsen during follow-up. This finding would have a significant impact on the current recommendations for treatment in patients with mitral regurgitation by supporting a conservative management approach.

DETAILED DESCRIPTION:
Current ACC/AHA guidelines recommend that patients with severe degenerative mitral regurgitation be considered for mitral valve surgery. There remains a debate within the cardiology community regarding the appropriate management of patients who remain asymptomatic. There are those who advocate for performing early "prophylactic" mitral valve surgery while others advocate clinical follow-up until triggers emerge with echocardiography historically being the method used for longitudinal assessment of cardiac anatomy and function. Two studies showed that only ~30% of asymptomatic severe mitral regurgitation made endpoints that triggered. However, these studies were limited and did not perform rigorous follow up assessment of regurgitant volume, left ventricular hemodynamics, exercise capacity, or quality of life assessment. In addition, in these studies mitral regurgitation and left ventricular size and function was assessed by echocardiography. Echocardiography has known limitations in assessing ventricular size and, as recent studies have shown, may not be the optimal modality to assess mitral regurgitant severity. MRI is the gold standard for non-invasive quantification of the left and right ventricles volumes and function and has emerged as a reference standard for quantifying mitral regurgitation. In this study the investigators will perform longitudinal follow-up data with cardiac MRI to inform the prophylactic surgery vs. close follow-up debate and to better define the natural history of this condition. The investigators hypothesize, that in the majority of patients mitral regurgitation will not worsen overtime, left ventricular hemodynamics will remain stable, exercise capacity will not decline, and symptoms will not worsen during follow-up. This finding would have a significant impact on the current recommendations for treatment in patients with mitral regurgitation by supporting a conservative management approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 yrs
2. able to give informed consent
3. Diagnoses of moderate or severe degenerative mitral regurgitation (based on the integrated approach recommended by the American Society of Echocardiography)

Exclusion Criteria:

1. Left ventricular ejection fraction <60%
2. Heart failure
3. Pulmonary hypertension (pulmonary artery systolic pressure >40mmHg at rest or >60mmHg with exercise as assessed by echocardiography)
4. Atrial fibrillation
5. Concomitant > mild aortic or mitral stenosis, >mild aortic or tricuspid or pulmonic regurgitation
6. Prior valvular heart disease surgery
7. Hypertrophic cardiomyopathy or an infiltrative cardiomyopathy
8. Unable to exercise on a treadmill
9. Symptomatic coronary artery disease
10. Comorbidities expected to impact functional capacity and confound symptom assessment (e.g COPD)
11. Expected lifespan of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with moderate or severe mitral regurgitation by echocardiography and remain asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in mitral regurgitant volume | Entry into study, 1 year, and 2 years
  Change in mitral regurgitant volume quantified by MRI over follow-up period

SECONDARY OUTCOMES:
Change in left ventricular end-diastolic volume | Entry into study, 1 year, and 2 years
  Change in left ventricular end-diastolic volume quantified by MRI over follow-up period
Change in symptoms and quality | Entry into study, 1 year, and 2 years
  Change in symptoms and quality of life as measured by EQ5DL questionnaires
Change in exercise capacity | Entry into study, 1 year, and 2 years
  Change in exercise capacity measured by treadmill exercise test
Follow up events | 1 yea, and 2 years
  Follow up events defined as death, need for surgery, heart failure symptoms, or valvular disease related hospitalizations
Change in degree of myocardial fibrosis | Entry into study, 1 year, and 2 years
  Change in degree of myocardial fibrosis measured as the percentage left ventricular hyperenhancement and change in mean ECV

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Uretsky S, Gillam LD, Biederman RWW, Han Y, Jacob R, Martin ET, Langer M, Choi AD, Sultan I, Cavalcante JL, Shah DJ, Tong MS, Wolff SD, Sakul S, Guglielmo M, Pontone G. Sex differences in pre- and post-surgical left ventricular remodelling and outcomes in primary mitral regurgitation. Eur Heart J Cardiovasc Imaging. 2025 Jul 31;26(8):1429-1437. doi: 10.1093/ehjci/jeaf151. PMID 40392571